CLINICAL TRIAL: NCT00797212
Title: Clinical Evaluation of the Apollo Blood Glucose Monitoring System With Alternative Site Testing [Commercial Name is CONTOUR® USB]
Brief Title: A New Glucose Meter With Alternative Site Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTD-2008-19
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Results first posted 2009-12-14 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subjects with diabetes (Other): Subjects with diabetes use a new Apollo Blood Glucose Monitoring System with blood obtained from the palm and forearm
  Interventions: Device: Apollo Blood Glucose Monitoring System

INTERVENTIONS:
Device: Apollo Blood Glucose Monitoring System — Subjects with diabetes use a new blood glucose monitoring system with blood taken from the palm and forearm. These blood glucose AST results are compared with results obtained by healthcare professionals (HCPs) from subject fingersticks.
  Other Names: Commercial name is CONTOUR® USB

SUMMARY:
The purpose of the study was to evaluate the performance of the blood glucose monitoring system when used with samples taken from the palm and forearm for alternative site testing (AST).

DETAILED DESCRIPTION:
The blood glucose monitoring system may be used for alternative site testing. The blood glucose results obtained by subjects with samples taken from the palm and forearm were compared with fingerstick capillary blood glucose results obtained from subjects by an HCP. Product labeling was evaluated for comprehension of performing alternative site testing as well as for additional meter features. User feedback about the system and its features was obtained.

ELIGIBILITY:
Inclusion Criteria:

* Have type 1 or type 2 diabetes
* Be >18<76 years of age at time of consent, with approximately 50% (+10%) being less than 55 years of age
* Be willing to complete all study procedures
* Be routinely testing their blood sugar at home (at least once per day)
* Be able to speak, read, and understand English and understand the Informed Consent document
* Be able to read the labeling instructions

Exclusion Criteria:

* Minors <18 years of age and adults >75 years of age
* Pregnancy
* Physical (dexterity), visual, or neurological impairments that would make the person unable to perform testing with the BGMS
* Disorders in the fingertip lancing areas
* Acute or chronic infections, particularly skin infections
* Infection with a blood borne pathogen
* Taking prescription anti-coagulants or having clotting problems that may prolong bleeding. Taking aspirin daily (81mg or 325 mg) is not reason for exclusion.
* Hemophilia or any other bleeding disorder
* Having a condition which, in the opinion of the Principal Investigator or designee, would put the person at risk or seriously compromise the integrity of the study
* Working for a competitive medical device company

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-11; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vimala Sethy, MD, PhD, Principal Investigator — Jasper Clinic, Inc.
Locations (1):
- Jasper Clinic, Inc., Kalamazoo, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects With Diabetes: Subjects with diabetes use a new blood glucose monitoring system with blood obtained from the palm and forearm.
Period: Overall Study
Arm/Group | Subjects With Diabetes
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Subjects With Diabetes
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 41
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 24
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of AST Results Within +/- 15mg/dL or +/- 20% of Fingerstick (FS)Blood Glucose Results
Description: Performance of the blood glucose monitoring system when the system is used for alternative site testing (AST) with samples from the palm and forearm compared with BGMS fingerstick capillary blood results obtained by an HCP
Time Frame: One hour
Population: per protocol
Measure: Number; unit: number of AST Blood Glucose Results
Arm/Group | Subjects With Diabetes
Number analyzed (Participants) | 50
number of AST Blood Glucose Results
  Results from palm (subject blood) (n=101) | 96
  Results from forearm (subject blood) (n=100) | 93

2. Secondary Outcome: Percentage of Participants Rated as <=3 (Labeling Comprehension)
Description: Study staff rated participants as to their success at performing meter testing. The rating scale was:
  1. Successful
  2. Successful after being referred to user instructions
  3. Successful with verbal assistance or review of part of user instructions (Similar to review of a specific function during a Customer Service call.)
  4. Unsuccessful (Incorrectly performed part of the testing regimen or required intervention by study staff.)
Time Frame: One hour
Population: per protocol
Measure: Number; unit: percent of participants
Arm/Group | Subjects With Diabetes
Number analyzed (Participants) | 50
percent of participants
  Fingerstick glucose result | 100
  Alternative site glucose result | 100

3. Secondary Outcome: Percentage of Participant Ratings for Overall Testing Experience With This Meter
Description: Subjects completed a questionnaire rating their overall experience with the Apollo Blood Glucose Monitor System (User feedback on the system). The rating scale was 0 (Unacceptable) to 4 (Excellent).
Time Frame: One hour
Population: per protocol
Measure: Number; unit: percent of participants
Arm/Group | Subjects With Diabetes
Number analyzed (Participants) | 50
percent of participants
  4 Excellent | 68
  3 Very Good | 26
  2 Good | 6
  1 Poor | 0
  0 Unacceptable | 0

ADVERSE EVENTS:
Arm/Group | Subjects With Diabetes
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less